CLINICAL TRIAL: NCT02243501
Title: Better Nights, Better Days: Improving Psychosocial Health Outcomes in Children With Behavioural Insomnia
Brief Title: Better Nights, Better Days for Typically Developing Children
Acronym: BNBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 228586
Record Dates: First submitted 2014-04-14; First posted 2014-09-18 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2018-12

CONDITIONS: Nonorganic Insomnia; Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The Intervention Group receives access to the BNBD intervention, and can access alternative resources while enrolled in the study. The BNBD intervention for caregivers of children 1 to 10 years with insomnia is a self-guided program delivered online. The intervention is conceptually consistent across age groups. Interactive and personalized content and evidence-based strategies are incorporated: sleep education, positive routines, faded bedtime with response cost, sleep restriction, extinction/graduated extinction, stimulus fading, and scheduled awakenings. BNBD includes five sessions available sequentially: Sleep Information; Healthy Sleep Practices; Settling to Sleep; Going Back to Sleep; Looking Back and Ahead. The completion time of the intervention will range from 5-10 weeks.
  Interventions: Behavioral: Intervention Group
- Usual Care Group (No Intervention): The Usual Care Group will receive no treatment until after the 8 month follow-up assessment. The Usual Care Group can access alternative resources and additional programs and services while enrolled in the study.

INTERVENTIONS:
Behavioral: Intervention Group — The BNBD intervention for caregivers of children 1 to 10 years with insomnia is a self-guided program delivered online. The intervention is conceptually consistent across age groups. Interactive and personalized content and evidence-based strategies are incorporated: sleep education, positive routines, faded bedtime with response cost, sleep restriction, extinction/graduated extinction, stimulus fading, and scheduled awakenings. BNBD includes five sessions available sequentially: Sleep Information; Healthy Sleep Practices; Settling to Sleep; Going Back to Sleep; Looking Back and Ahead. The completion time of the intervention will range from 5-10 weeks.
  Other Names: Better Nights, Better Days
  Arms: Intervention Group

SUMMARY:
Up to 25% of children suffer from sleep problems categorized as "insomnia": difficulty settling, falling asleep, and staying asleep. This leads to daytime sleepiness and negatively effects behaviour, mood, and academic performance. It also has negative effects on primary caregiver's sleep and their daytime functioning. Despite robust evidence supporting the efficacy of behavioural treatments for insomnia in children, very few receive these treatments. The most common treatment for insomnia in children is medication. This pattern of care is troubling because there are no approved medications for insomnia in children, and there are concerns about the safety and side effects of these medications. One of the primary reasons for the low rate of evidence-based treatment is the shortage of available treatment resources for both parents and health care providers.

When evidence-based treatments are available, they are usually provided in a traditional service delivery framework. These traditional approaches are often very difficult for parents to access due to scheduling conflicts, incidental costs, and travel difficulties. Thus, there is a critical need for access to effective interventions focused on insomnia for children, and increased knowledge for parents and health care providers about appropriate treatments for insomnia.

The Better Nights, Better Days (BNBD) program will provide a potential solution to one of the most common treatment barriers: access to care. BNBD will provide a readily accessible distance treatment via the internet, to increase access to evidence-based care for insomnia in typically developing children aged 1 to 10. BNBD was developed based on evidence-based programs and extant literature. The investigators will conduct a randomized controlled trial (RCT) in which participants (primary caregivers of children ages 1 to 10 years with insomnia) will be assigned to Intervention or Usual Care based on a 1-to-1 allocation. The effects of this behavioural sleep intervention will be assessed at 4 and 8 months post baseline assessment. Assessment will include both sleep and daytime functioning of the children, and daytime functioning of their caregivers.

This study aligns with the recognized need to more rapidly transfer new scientific knowledge to improve patient care and population health, and targets the validation of new treatment delivery models to increase availability of effective treatment.

DETAILED DESCRIPTION:
Rationale:

Evidence demonstrates that behavioural interventions should be the first line of treatment for children with insomnia, but this is not typically the case. Evidence-based behavioural intervention protocols are not readily available for clinical use, and their lack of implementation indicates inadequate knowledge translation. When evidence-based treatments are available, they are usually provided in a traditional service delivery framework (i.e., face-to-face therapy, small group therapy). These traditional approaches are often very difficult for parents to access due to scheduling conflicts, incidental costs, and travel difficulties. Thus, there is a critical need for access to effective interventions focused on insomnia for children, and increased knowledge for parents and health care providers about appropriate treatments for insomnia. The Better Nights, Better Days (BNBD) program will bridge this gap as we will provide a potential solution to one of the most common treatment barriers, access to care.

Intervention:

The BNBD intervention for children aged 1 to 10 years with insomnia is a bilingual, self-guided program delivered online. The intervention incorporates evidence-based strategies, including sleep education, positive routines, faded bedtime with response cost, sleep restriction, extinction/graduated extinction, stimulus fading, and scheduled awakenings. The intervention is comprised of five sessions made available sequentially to participants. The completion time of the intervention will range from 5-10 weeks. Each session will provide factual information to parents, strategies for implementation of best practices to address sleep problems, and access to additional help and advice. There is also a "Reward Centre" where parents can learn how to use reinforcement for children (e.g., sticker charts) to help support the implementation of these sleep intervention strategies. Participants complete a short Sleep Diary for a minimum of 5 days for each session throughout this intervention so that they can receive feedback on their progress. The intervention delivers the interactive, personalized cognitive and behavioural change strategies accessed through participants' desktops, laptops, tablets and smartphones. The program can be used at a time that is convenient for the participants, removing barriers to care and providing services in the comfort and privacy of their own homes.

Objectives and Hypotheses:

The study will evaluate the effectiveness of the BNBD online intervention for insomnia in children 1-10 years of age. The primary objective is to assess the immediate impact (Baseline vs. 4 month) of the intervention on children's sleep. The two hypotheses for the primary outcomes are:

1. Improvements in sleep efficiency calculated using actigraphy data in the Intervention Group compared with the Usual Care Group, and
2. Improvements in sleep efficiency calculated using Sleep Diary data in the Intervention Group compared with the Usual Care Group

The secondary objectives are: a) to evaluate the longer-term impact (baseline, 4, 8 months) on children's sleep and psychosocial health and, b) to examine the impact on parent daytime fatigue and psychosocial health outcomes. The four hypotheses of the secondary outcomes are:

1. Children in the Intervention Group will show improvement compared to children in the Usual Care Group at the two follow-up time points in their symptoms of insomnia based on improvements in sleep efficiency calculated using actigraphy and Sleep Diary data in the Intervention group compared with the Usual Care group.
2. Children in the Intervention Group will show improvement compared to children in the Usual Care Group at the two follow-up time points in their symptoms of insomnia based on the total score from the Behavioural Insomnia Questionnaire (BIQ) and Tayside Children's Sleep Questionnaire (TCSQ; toddler and pre-schoolers) / Sleep Disturbance Scale for Children (SDSC; school-age).
3. Children in the Intervention group, compared to children in the Usual Care Group, will show improved psychosocial health based on the internalizing and externalizing total scores from the Child Behaviour Checklist (CBCL/1 ½-5 and CBCL/6-18) and the total score from the Pediatric Quality of Life (Peds- QL).
4. Parents randomized to the Intervention Group, compared to parents randomized to the Usual Care group, will show at all follow-up time points:

1.Decreased daytime fatigue based on the Single Item Fatigue Impact Scale (SIFIS) 2.Improved psychosocial health as assessed by the total score of the Depression, Anxiety and Stress Scales (DASS-21) 3.Improved parenting strategies as assessed by the total score of the Parenting Scale (PS)

Exploratory analyses will examine age effects, the impact of the intervention on children's physical health, as well as process-level evaluation and implementation questions, exploring how BNBD works (e.g., changes in specific sleep behaviours such as bedtime routines, and predictors of treatment success).

Study Design:

The study is a two-arm Randomized Controlled Tiral (RCT) design, using 1-to-1 allocation, comparing participants assigned to receive either the BNBD online program for parents (Intervention Group) or the control group (Usual Care Group) who will not receive the intervention. The intervention will be delivered across Canada. The study will be coordinated through Corkum LABS at Dalhousie University.

Randomization will be used to minimize bias in the assignment of participants to either group, to increase the likelihood that known and unknown participant attributes (e.g., demographic and baseline characteristics) are evenly balanced, and to enhance the validity of statistical comparisons across groups.

Participants will be stratified at randomization by three age groups (Toddler, Pre-School, School-Aged) and two primary languages (English and French). Targets will be set for each variable - 1/3 of sample in each age group and 20% of sample French speaking, modelling the Canadian populatipm. This will ensure the study population is representative and balanced. Within each stratum, subjects will be randomized using an equal allocation ratio of 1:1. Both the Intervention Group and Usual Care Group will be able to access alternative resources and additional programs and services while enrolled in the study.

Blocks of 6 will be used to randomize the participants for each strata. The block size is short enough to prevent imbalance, and long enough to prevent guessing allocation in trials.

The power analyses indicate the need to have 250 participants in total who complete the final follow-up assessment at 8 months post randomization. Based on the Investigators past intervention research as well as sleep intervention trials in the literature, 500 participants who have successfully completed eligibility will be needed using an estimated 50% drop out rate from post-eligibility to the final follow-up assessment at 8 months. More specifically, loss of participants at each stage is estimated to be the following: 22% from post eligibility to end of baseline, 15% from post-randomization to 4 month assessment, and 13% from the 4 month to 8 month assessment.

Outcome measures will be administered to all participants at Baseline and at 4 and 8 months post-randomization online through the REDCap database. Data collected at 8 months will assess the degree of maintenance of any initial treatment effects on children's sleep in each age group, as well as examine the longer-term impact of the intervention on child and parent psychosocial health. The REDCap database will automatically contact participants via email to complete assessments. There will be automated emails from REDCap followed by phone calls from the research staff to ensure that outcome data is collected.

Study participation ends for participants in both study groups after completing the 8 month follow-up assessment. Participants in the Usual Care group will gain access to the BNBD program after their study participation is complete. The BNBD program will be accessible for the Usual Care group for 3 months.

Subject Population:

A total of 500 participants will be eligible to participate in the study. Participants will be recruited from across all Canadian provinces and territories. A target of 100 English-speaking participants will be recruited from across four geographical regions of Canada (Atlantic, Central, Prairies, West Coast and Northern Territories).

Data Analysis:

The primary outcome measures that will be used to evaluate the impact of the intervention program on insomnia symptoms are sleep efficiency based on actigraphy data and sleep efficiency based on Sleep Diary data. Two primary outcome measures are included in order to capture the variables of interest using both an objective measure of sleep (i.e., actigraphy) and a parent-report/subjective measure of sleep (i.e., Sleep Diary), thus allowing for comparison with existing research in the field. Another reason for using both objective and subjective measures is that it has been found that unblinded RCTs (i.e., in which participants know their group assignment such as the current study) have been demonstrated to be biased in favour of the active treatment, and it has been suggested that an objective measure (e.g., actigraphy) should be utilized in the assessment of outcomes. Secondary outcomes will examine the longer-term impact of change in sleep as well as the impact on the child's psychosocial health (behavioural, attentional, and emotional functioning) over the duration of the 8 month trial. We will also examine the impact on parents' fatigue levels and psychosocial health.

Primary Outcome: A mixed effect General Linear Models will be fit to the data to test if the Intervention group demonstrates improved outcomes compared to the Usual Care group. The dependent variables will be the primary outcomes assessed at 4 and 8 months post-randomization (sleep efficiency on actigraphy and the Sleep Diary). Participants will be modelled as random effects group (Intervention vs. Usual Care) and baseline covariates (age and language) will be modelled as fixed effects. A significant interaction effect between time (baseline, 4 and 8 month) and group will indicate an intervention effect for treatment.

Secondary Outcome: All secondary outcomes will be separately analyzed using Hierarchical Linear Modelling and will test differences between the two groups (Intervention vs. Usual Care) in the growth curves modelling changes in the outcome variables across the four points of measurement, controlling for age, language and other covariates.

Exploratory analyses: The investigators will examine the possibility of differential response to treatment across the three age groups using growth curve modelling of the two primary outcomes (actigraphy and Sleep Diary).

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet the following criteria to be eligible to participate in the study:

1. Primary caregiver of a child aged 1 to 10 years.
2. Live in any province or territory in Canada.
3. Have regular access to high speed internet connection and an email account.
4. Comfortable communicating in English or French for day-to-day tasks (e.g., listening to the news on the radio or watching TV, reading books, magazines, etc.).
5. Child has insomnia, defined as having Sleep Onset Disturbance. For Sleep Onset Disturbance, child must meet two of the following three criteria. These episodes must have been occurring for at least one month:

1. More than three reunions for 12-24 month olds/more than two reunions for >24 month olds that occur two or more nights per week 2. 30 or more minutes to fall asleep for 12-24 month olds/20 or more minutes to fall asleep for >24 month olds 3. Parent remains in room for sleep onset for two or more nights per week

Exclusion Criteria:

Potential participants who meet any of the following criteria are not eligible to participate in the study:

1. Parent wishes to "bed-share" with his/her child.
2. Child has a probable intrinsic sleep disorder (e.g., sleep apnea) as assessed using the Pediatric Sleep Questionnaire (PSQ).
3. Child has a significant medical disorder that interferes with sleep (e.g., asthma attacks during night, tube feeding, non-ambulatory, severe developmental disability affecting sensory systems such as vision).
4. Child has a mental health disorder that has required hospitalization or residential care and/or current use of psychotropic medications which are known to interfere with sleep (e.g., stimulant medication for ADHD).

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 534 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Efficiency and Onset Latency from Baseline to 8 Month Follow-up with Actigraphy | 8 months
  Actigraphy involves measurement of motor activity using an accelerometer-based, battery-operated device. The investigators will use actigraphy to collect information about changes in children's sleep efficiency (captured from lights out to awakening), sleep onset, total sleep time, and night wakings from baseline to 4 month and 8 month follow-up. Actigraphy data have been shown to be highly concordant with polysomnographic (PSG) data for identifying sleep and waking (85-90%) and to distinguish effectively between sleep-disturbed children and controls. The investigators will use Philps Respironics Actiwatch 2 actigraphs. Actigraphy data will be collected for a one week period at baseline, and 4 months and 8 months post randomization. Participants are instructed to ensure their child wears their actigraph during the 7 days of Sleep Diary collection.
Change in Sleep Efficiency and Onset Latency from Baseline to 8 Month Follow-up with Sleep Diary | 8 months
  Sleep Diaries will be used to document sleep variables over a number of days/nights. A composite score will capture bedtime resistance, difficulties falling asleep and night wakings, as these are the key features of insomnia in children. Parents record information about their children's sleep and sleep behaviours for a one week. The Sleep Diary contains 25 items specifically measuring; sleep duration, night time sleep duration, daytime sleep duration, sleep onset latency, bedtime, wake time, presence and frequency of night awakening, and the presence and frequency of bedtime resistance. Sleep Diaries also provide a measure of time spent in bed extracted from the time the light was turned off ("Down for the night") to the time lights were turned on ("Up for the day"). Sleep Diaries are administered to participants at the 3 assessment periods to assess change over baseline to 4 month and 8 month follow-up. Sleep diaries have demonstrated good face validity and high internal consistency.

SECONDARY OUTCOMES:
Tayside Children's Sleep Questionnaire (TCSQ) | 8 months
  Two questionnaires will be used to assess children's sleep / insomnia, depending on the age of the child, at baseline, 4 month and 8 month assessment periods. The Tayside Children's Sleep Questionnaire (TCSQ) consists of 10 items and will be used to measure insomnia symptoms in children aged 1-5 years. Only the first 9 items are used for scoring, and the last item is included to assess how parents view their child's sleep problem, but is excluded from data analysis. The TCSQ has been validated for its use to accurately measure sleep problems.
Pediatric Quality of Life (Peds-QL) | 8 months
  The Pediatric Quality of Life (Peds-QL) questionnaire is used to assess children's physical and psychosocial health at baseline, 4 month and 8 month assessment periods. The participant will complete the form for ages 2-4, 5-7, or 8-12. The Peds-QL is a validated, 23-item modular tool designed to measure health related quality of life (HRQoL) in children and adolescents across 4 domains: physical, emotion, social and school functioning. The questionnaire uses a Likert Scale anchored 0 "never" to 4 "almost always", with reverse-scored answers linearly transformed to a 0-100 scale, with higher scores reflecting higher health related quality of life. The cut-off score assigned to physical health is any value 1 SD below the population sample mean, and this is also applied to psychosocial health.
Child Behaviour Checklist (CBCL) | 8 months
  The Child Behavior Checklist (CBCL) for ages 1 ½-5 and 6-18 will be used to assess the child's daytime functioning and psychosocial health at the three assessment periods. CBCL/1 ½-5 responses are scored and summed across subscales (Emotionally Reactive, Anxious/Depressed, Somatic Complaints, Withdrawn, Sleep Problems, Attention Problems, Aggressive Behaviour), combined into "internalizing" and "externalizing", and compared to a normative sample indicating the child's behaviour falling within "normal" limits, "borderline clinical", or "clinical". CBCL/6-18 responses are scored and summed across subscales (Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-breaking Behaviour and Aggressive Behaviour), grouped into either internalizing or externalizing factors with total scores, compared to a normative sample indicating where the child's behaviour falls. The CBCL is psychometrically sound.
Teacher Report Form (TRF) | 8 months
  The Caregiver Teacher Report Form (C-TRF) for children 1 ½ to 5 and Teacher Report Form (TRF) 6-18 is used to assess children's daytime functioning and psychosocial health, obtained from an informant to validate parent reports. The forms received by teachers are dependent on the child's age. The TRF measures a child's adaptive functioning and behavioural problems with 100 items on a 3-point Likert-scale anchored from 0 "not true" to 2 "very true or often true", with the added textboxes for qualitative feedback. Both TRFs are optional measures that participants may forward to their child's teachers, and are administered at baseline, 4 months and 8-months follow up. The TRF has demonstrated good psychometric properties, high test-retest reliability and internal consistency.
Single Item Fatigue Impact Scale (SIFIS) | 8 months
  The SIFIS is a single item that measures the severity of fatigue on caregivers. Responses are recorded on a Likert-scale anchored from 0 "none" to 10 "a severely disabling effect". Participants receive the SIFIS at baseline, 4 and 8 month assessment periods. The SIFIS was adapted from Chan and colleagues' (2003) 40-item Fatigue Impact Scale, a measure with sound psychometric properties, demonstrating high internal consistency and the adequate correlations between each item's rating and the summed ordinal ratings of the remaining items, high construct validity and responsiveness.
Depression Anxiety Stress Scale (DASS-21) | 8 months
  The Depression Anxiety and Stress Scale (DASS-21) is used to measure self-reported parent distress. Using 21 items, participants indicate to what extent they have experienced certain mental health disorder symptoms in the past month. Items are anchored from 0 "did not apply to me at all" to 3 "applied to me very much or most of the time. Responses are scored into three subscales: depression, anxiety and stress. These subscales are combined to obtain a measure of general stress, which is the variable that used in this study. The DASS-21 has been validated for its use to measure parent distress in a community, nonclinical sample with strong internal consistency. Concurrent validity was also validated, and the DASS-21 also demonstrates high sensitivity to effects of parent-focused interventions.
Parenting Scale (PS) | 8 months
  The Parenting Scale (PS) is used to measure dysfunctional parenting practices consisting of 30 items. This rating scale was designed to measure dysfunctional parenting across three stable factors; laxness, over reactivity, and verbosity. Participants are instructed to select a circle on a visual analogue scale to identify to what extent they engage in certain parenting practices (e.g. giving child several reminders/warnings as opposed to one reminder/warning). The measure has established test reliability and validity.
Sleep Disturbance Scale for Children (SDSC) | 8 months
  Two questionnaires will be used to assess children's sleep / insomnia, depending on the age of the child, at baseline, 4 month and 8 month assessment periods. The Sleep Disturbance Scale for Children (SDSC) will be used to measure insomnia in children aged 6-10. The SDSC will be used to measure initiation and maintenance of sleep. The SDSC has been validated with high sensitivity specificity, and reliability coefficients.

OTHER OUTCOMES:
Demographic Questionnaire (DQ) | 8 months
  A Demographic Questionnaire (DQ) is used to collect basic demographic information of the participant, the spouse/partner of the participant (if applicable), and the child of the participant. 29 items were compiled from the format of the Canadian Consensus, and the National Longitudinal Survey of Children and Youth (2011). Questions pertain to the age, sex, number of adults living in the home, relationship to the child participating, marital status, ethnic or cultural heritage, highest level of education completed, employment status, work hours, job position, household income, if their spouse/partner live in their home (if applicable), and their spouse/partner's relationship with the participants' child. If applicable, the same questions are asked about the caregiver's spouse/partner and their child. The information collected will be used to describe the sample and will allow us to determine the representativeness of the sample to the Canadian population.
Children's Physical Activity Index (PAI) | 8 months
  The Children's Physical Activity Index CPAI is adapted from the Children's Physical Activity Questionnaire from the Canadian Health Measures Survey (2007) and is used to measure the child's physical activity levels. Participants will receive the CPAI at baseline and 8 month follow-up. When the CPAI is administered, participants will be asked to provide responses to questions aimed at understanding the child's levels of activity and/or inactivity. Response options vary from 5-8 options given, ranging from "never" engaging in a particular activity (either related to activity or inactivity) or "always".
Body Mass Index (BMI) | 8 months
  Body Mass Index (BMI) is collected to determine the physical fitness of the child. BMI will be calculated using The Dieticians of Canada BMI calculator (2015) for children and teens. After the BMI is calculated, percentile charts are calculated. BMI is measured at baseline and 8 month follow-up. Participants are instructed to use a measuring tape and scale to obtain accurate measurements for the height, weight and waist circumference of their child. Participants then provide the exact height, weight, waist circumference, and BMI score. Reference for these instructions were adapted from The Dieticians of Canada BMI calculator website (2015).
Parenting Rating of Clinical Significant Improvement (PRCSI) | 8 months
  The Parents Rating of Clinically Significant Improvement (PRCSI) is used to assess parents' percentage of satisfaction with the intervention progress. The PRCSI was adapted from Montgomery, Stores and Wiggs (2004) to be appropriate for measuring clinically significant improvement using analogue scale self-reports. The PRCSI contains 3 items requiring parents to use an analogue scale to record their satisfaction responses and is administered at baseline, 4 month and 8 month follow-up. This measure is also completed by parents in the Intervention Group prior to each intervention session.
Treatment Utilization (TU) | 4 months
  The Treatment Utilization (TU) questionnaire was adapted from The Parenting Matters Program. It measures the extent to which parents utilize treatment resources (i.e. family physicians). This is a predictor of treatment success and the responses is used to assess the need for treatment intervention. The TU includes 27 items divided into 8 item categories: family physician, pediatrician, other person or place for regular health care, urgent care and emergency room, specialized health services, cost, medications, and other sources of help or advice. The TU is administered at the baseline, 4 and 8 month follow-up.
Willingness to Pay (WP) | 4 months
  The Willingness to Pay (WP) questionnaire will be used to assess participants' perceptions of the value of the program. The WP is administered at baseline and only administered to those in the Intervention Group at 4 month follow-up.
Barriers to Treatment Participation Scale (BTPS) | 4 months
  The Barriers to Treatment Participation Scale (BTPS) is a 12 item questionnaire used to assess participants' experience of obstacles or barriers to participating in their children's treatment, treatment demands or issues, and perceived relevance of treatment. Items are anchored on a 5-point Likert-scale that ranges from 1 "never a problem" to 5 "very often a problem". Previous studies have demonstrated adequate internal consistency reliability. The BTPS will be administered to the Intervention Group at the 4 month follow-up.
Client Satisfaction Questionnaire (CSQ-8) | 4 months
  The Client Satisfaction Questionnaire (CSQ-8) is used to measure participant satisfaction with the BNBD intervention. The CSQ-8 is an 8 item measure that is widely used in primary care and mental health treatment and measures satisfaction using a 4-point Likert-scale ranging from 1 being "No, definitely not" to 4 "yes, definitely" in terms of the participant satisfaction. The CSQ-8 is administered to participants receiving the intervention at 4 months follow-up. An overall score for the CQS-8 is produced by summing all item responses producing scores ranging from 8 to 32, with higher values indicating higher satisfaction. The CSQ-8 is a well-established measure for satisfaction with an established internal consistency.
Readiness for Change (RC) | Baseline
  The Readiness for Change (RC) questionnaire assesses whether participants are mindful and willing to adjust their parenting practices. This is used as a predictor of treatment engagement. Several studies have utilized the RC measure in the context of parenting successfully to predict parent commitment to treatment. Participants are instructed to record their responses on a 6-point scale ranging from "strongly disagree" to "strongly agree" with the option to also provide the response "does not apply". The RC is administered at baseline.
Bedtime Routines Questionnaire (BRQ | 4 months
  The Bedtime Routines Questionnaire (BRQ) is used to measure bedtime routine activities using 31 items. This questionnaire provides information about how the participants' child goes to bed during weekdays and weekends. Responses are measured on a 5-point frequency scale ranging from 1 "almost never" to 5 "nearly always". BRQ responses are good predictors for treatment outcome, and increased agreement with the use of limit setting strategies and rewards related to better outcomes in the child's sleep. The BRQ has demonstrated strong psychometric properties. It has an acceptable to excellent internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Penny V Corkum, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corkum PV, Reid GJ, Hall WA, Godbout R, Stremler R, Weiss SK, Gruber R, Witmans M, Chambers CT, Begum EA, Andreou P, Rigney G. Evaluation of an Internet-Based Behavioral Intervention to Improve Psychosocial Health Outcomes in Children With Insomnia (Better Nights, Better Days): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Mar 26;7(3):e76. doi: 10.2196/resprot.8348. PMID 29581089